CLINICAL TRIAL: NCT01002807
Title: Bioavailability Study of Two Prototype Fixed Dose Combination (FDC) Formulations of 10 mg Dapagliflozin and 1000 mg Metformin Extended Release (XR) Tablet Relative to Dapagliflozin 10 mg Tablet and Glucophage® XR 2 X 500 mg Tablets Coadministered to Healthy Subjects in a Fasted State
Brief Title: Bioavailability Study of Fixed Dose Combination (FDC) Formulations of Dapagliflozin and Metformin XR Versus Individual Component Coadministered to Healthy Subjects in a Fasted State
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: MB102-065
Record Dates: First submitted 2009-10-26; First posted 2009-10-27 (Estimated); Last update posted 2016-10-17 (Estimated); Status verified 2016-10

CONDITIONS: Type 2 Diabetes Mellitus (T2DM)
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dapagliflozin; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- FDC of dapagliflozin/metformin XR (Other)
  Interventions: Drug: Dapagliflozin; Drug: Metformin XR
- FDC of dapagliflozin/reduced mass metformin XR (Other)
  Interventions: Drug: Dapagliflozin; Drug: Metformin XR
- dapagliflozin and Glucophage® XR (Other)
  Interventions: Drug: Dapagliflozin; Drug: Glucophage

INTERVENTIONS:
Drug: Dapagliflozin — Tablets, Oral, 10 mg, Single Dose
Drug: Metformin XR — Tablets, Oral, 1000 mg, Single Dose
  Arms: FDC of dapagliflozin/metformin XR; FDC of dapagliflozin/reduced mass metformin XR
Drug: Glucophage — Tablets, Oral, 1000 mg, Single Dose
  Other Names: Glucophage™
  Arms: dapagliflozin and Glucophage® XR

SUMMARY:
To assess the relative bioavailability of dapagliflozin and metformin from the two FDC formulations, comprised of 10 mg dapagliflozin and 1000 mg metformin XR, relative to coadministration of a dapagliflozin 10 mg tablet and 2 x 500 mg Glucophage® XR tablets, in healthy subjects in a fasted state.

ELIGIBILITY:
Inclusion Criteria:

* Men and women ages 18 to 45 inclusive
* Healthy subjects as determined by no clinically significant deviation from normal in medical history, physical examination, ECGs, and clinical laboratory determinations
* Body Mass Index (BMI) of 18 to 32 kg/m2, inclusive. BMI = weight (kg)/ [height (m)]2

Exclusion Criteria:

* WOCBP who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period and for up to 8 weeks after the last dose of investigational product
* Any significant acute or chronic medical illness
* Current or recent (within 3 months) gastrointestinal disease
* Any major surgery within 4 weeks of study drug administration
* Glucosuria at screening
* Abnormal liver functions tests (ALT, AST or total bilirubin > 10% above ULN)
* Presence of edema on physical exam
* History of diabetes mellitus
* History of heart failure
* History of renal insufficiency
* History of chronic or recurrent UTI (defined as 3 occurrences per year) or UTI in the past 3 months
* History of recurrent (defined as 3 occurrences per year) or recent vulvovaginal mycotic infections
* Estimated creatinine clearance (ClCR) of < 80 mL/min using the Cockcroft Gault formula
* History of allergy or intolerance to metformin or other similar agents

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2009-11; Primary Completion 2009-12 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Blood samples to measure the pharmacokinetic parameters Cmax and AUC for the combination products versus each investigational product alone | 48 hours post-dose

SECONDARY OUTCOMES:
Safety and tolerability measures (adverse events, physical exams, vital signs, ECGs, and clinical laboratory assessments) | 15 timepoints in 48 hours time interval

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Ppd Development, Lp, Austin, Texas, United States

REFERENCES:
- See also: MB102-065_redacted_CSR_synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=3650&filename=MB102-065_redacted_CSR_synopsis.pdf